CLINICAL TRIAL: NCT06998134
Title: Toward Ubiquitous Lower Limb Exoskeleton Use in Children and Young Adults: Exploratory Observational Analysis of Novel Robotic Control Strategies
Brief Title: Toward Ubiquitous Lower Limb Exoskeleton Use in Children and Young Adults
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10002278; 002278-CC
Record Dates: First submitted 2025-05-30; First posted 2025-05-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-30

CONDITIONS: Muscle Weakness; Problems Moving Their Arms and Legs
Keywords: Cerebral Palsy (CP); muscular dystrophy (MD); Spina Bifida; incomplete spinal cord injury
MeSH Terms: conditions — Muscle Weakness; Cerebral Palsy; Muscular Dystrophies; Spinal Dysraphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cerebral Palsy (CP): Male and female age 5-25
  Interventions: Device: Extension assist knee ankle foot orthosis (EA-KAFO)
- Incomplete Spinal Cord Injury: Male and female age 5-25
  Interventions: Device: Extension assist knee ankle foot orthosis (EA-KAFO)
- Muscular Dystrophy: Male and female age 5-25
  Interventions: Device: Extension assist knee ankle foot orthosis (EA-KAFO)
- Spina Bifida: Male and female age 5-25
  Interventions: Device: Extension assist knee ankle foot orthosis (EA-KAFO)

INTERVENTIONS:
Device: Extension assist knee ankle foot orthosis (EA-KAFO) — A lower limb exoskeleton that has one actuated degree of freedom at the knee (flexion/extension) and a passive degree of freedom at the ankle (plantar/dorsiflexion).

SUMMARY:
People with cerebral palsy (CP), muscular dystrophy (MD), spina bifida, or spinal cord injury often have muscle weakness, and problems moving their arms and legs. The NIH designed a new brace device, called an exoskeleton, that is worn on the legs and helps people walk. This study is investigating new ways the exoskeleton can be used in multiple settings while performing different walking or movement tasks, which we call ubiquitous use. For example, we will ask you to walk on a treadmill at different speeds, walk up and down a ramp, or walk through an obstacle course. Optionally, the exoskeletons may also use functional electrical stimulation (FES), a system that sends electrical pulses to the muscle to help it move the limb.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

The following exploratory observational study is designed to create a framework that permits rapid development, piloting, and acute evaluation of pediatric exoskeleton control paradigms for daily, ubiquitous use across multiple settings. Most existing evaluations of pediatric exoskeleton control modes are limited to a flat walking task.The novelty of this study design is the translation of control modes to different functional tasks and comparisons between fixed and adaptive parameters across the tasks. Across all participants, three main control modes will be tested: assist, resist, and interleaved (alternating assist and resist). Control parameters will either be fixed for all tasks conducted or may adapt based on the motions of a given activity. Following informed consent and assent, screening, and calibration of control parameters, an acclimation period to the exoskeleton and control modes will occur. Each control mode will be tested across ubiquitous activities of daily living and outcomes will be compared to baseline (without wearing the exoskeleton). Our central hypothesis is that existing control paradigms that have been previously validated in walking can be successfully translated to improve knee extension deficiency and/or knee extensor muscle activity in multiple different functional mobility tasks.

OBJECTIVES:

* Primary Objectives: 1) To evaluate acute biomechanical and neuromuscular effects of pediatric exoskeleton control paradigms on knee extension deficiency across ubiquitous tasks and 2) Assess whether controller behavior and performance align with the intent of its prescribed design consistently across tasks.
* Secondary objectives: 1) Measuring functional performance of tasks conducted with each control paradigm and 2) Characterizing muscle activation of knee extensors during each task.

ENDPOINTS:

Primary Endpoints:

* To evaluate knee extension deficiency, we will use 1) Peak knee extension and 2) Range of knee angle excursion (difference between maximum extension and flexion). These endpoints will be measured and compared between each control strategy within each task during the assessment visit.
* To characterize controller behavior and performance, we will use the root mean square error (RMSE) between the exoskeleton knee torque profile delivered in real-time and the ideal knee torque profile computed from the user s kinematics. This endpoint will be measured during each assessment visit.

Secondary Endpoints:

-To evaluate functional performance in:

* self-selected speed treadmill walking, overground walking, stairs, and ramps, we will use gait speed, stride length, and number of gait cycles.
* variable-speed treadmill walking, we will use cadence, stride length, and number of gait cycles.
* Timed Up and Go and stairs, we will use the duration of the task.
* the Standardized Walking Obstacle Course, we will use the time to traverse the environment.
* the 6-Minute Walk Test, we will use the distance covered during the task.
* the squat test, we will use the number of squats completed.

These endpoints will be measured and compared between each control strategy used within each task during the assessment visit.

To characterize muscle activation, we will use 1) peak knee extensor activation during the task and 2) area under the normalized EMG curve over the duration of the task. These endpoints will be measured and compared between each control strategy used within each task during the assessment visit.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated separate informed consent and assent forms for screening purposes. Upon inclusion in the protocol, provision of signed and dated informed consent and assent forms to begin participation in the study will be necessary.
* Stated willingness to comply with all study procedures and availability for the duration of the study, or alternatively, ability to do so based on parent report and physician observation during history and physical examination.
* Age 5 to 25 years old. Importantly, we included young adults (18-25 years old) because longterm outcomes for adults with cerebral palsy include loss of ambulatory ability. While studies of conventional gait training in this population have been conducted, use of exoskeletons in this population is very limited. Given the potential benefit of exoskeletons to reduce knee extension deficiency, it is important to determine whether novel controllers we develop are also tolerated and effective in this age group.
* Either has a gait pathology arising from a diagnosis of CP, MD, SB, or iSCI or has no gait pathology.
* Knee joint range of motion of at least 25 degrees in the sagittal plane (knee extension/flexion) assessed with the hip extended in a supine position. Hamstring contracture as assessed by the straight leg raising test does not limit ability to participate in the study.
* Ankle joint range of motion of at least 15 degrees in the sagittal plane (dorsi-plantarflexion) with the foot in neutral alignment.
* Able to walk at least 10 feet without stopping with or without a walking aid.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any neurological, musculoskeletal, or cardiorespiratory injury, health condition, or diagnosis other than CP, MD, SB, or iSCI that would affect the ability to walk as directed with the robotic exoskeleton.
* A history of uncontrolled seizures in the past year.
* Pregnancy based on self-reporting. We excluded pregnancy due to confounding factors of pregnancy on gait.
* Adult unable to consent for themselves at screening visit.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient age 5-25 cerebral palsy (CP), muscular dystrophy (MD), spina bifida, or spinal cord injury often have muscle weakness, and problems moving their arms and legs
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-08-18 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Evaluate acute biomechanical and neuromuscular effects of pediatric exoskeleton control paradigms on knee extension deficiency across ubiquitous tasks. | 4 months
  To evaluate knee extension deficiency, we will use:1) Peak knee extension and2) Range of knee angle excursion (difference between maximum extension and flexion).These endpoints will be measured and compared between each control strategy within each task during the assessment visit.

SECONDARY OUTCOMES:
Assess whether controller behavior and performance align with the intent of its prescribed design consistently across tasks. | 4 months
  To ensure controllers are appropriately developed for ubiquitous use, it is vital to determine whether their intended behavior is consistent with design specifications across tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Bulea, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hirtz D, Thurman DJ, Gwinn-Hardy K, Mohamed M, Chaudhuri AR, Zalutsky R. How common are the "common" neurologic disorders? Neurology. 2007 Jan 30;68(5):326-37. doi: 10.1212/01.wnl.0000252807.38124.a3. PMID 17261678
- [Background] Emery AE. The muscular dystrophies. Lancet. 2002 Feb 23;359(9307):687-95. doi: 10.1016/S0140-6736(02)07815-7. PMID 11879882
- [Background] Mitchell LE, Adzick NS, Melchionne J, Pasquariello PS, Sutton LN, Whitehead AS. Spina bifida. Lancet. 2004 Nov 20-26;364(9448):1885-95. doi: 10.1016/S0140-6736(04)17445-X. PMID 15555669
- [Background] McDonald JW, Sadowsky C. Spinal-cord injury. Lancet. 2002 Feb 2;359(9304):417-25. doi: 10.1016/S0140-6736(02)07603-1. PMID 11844532
- [Background] Damiano DL, Abel MF. Relation of gait analysis to gross motor function in cerebral palsy. Dev Med Child Neurol. 1996 May;38(5):389-96. doi: 10.1111/j.1469-8749.1996.tb15097.x. PMID 8698147
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002278-CC.html